CLINICAL TRIAL: NCT06446310
Title: A Randomised, Double-Blind, Placebo-Controlled, Multicentre, Phase 3, Clinical Study of QLG2198 in Haemodialysis Adult Subjects With Moderate-to-Severe Pruritus
Brief Title: Phase 3 Study of QLG2198 in Haemodialysis Chinese Adult Subjects With Moderate-to-Severe Pruritus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical (Hainan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLG2198-301
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Uremic Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 12-weeks double-blind period-QLG2198 (Experimental): Interventions:
  Drug: QLG2198 Injection
  Interventions: Drug: QLG2198
- 12-weeks double-blind period- placebo (Placebo Comparator): Interventions:
  Drug: Placebo Injection
  Interventions: Drug: Placebo
- 14-weeks open-label period following the double-blind period- QLG2198 (Experimental): Interventions:
  Drug: QLG2198 Injection
  Interventions: Drug: QLG2198

INTERVENTIONS:
Drug: QLG2198 — Participants receive QLG2198 three times a week (0,5 micrograms/kg dry body weight). QLG21988 is administered by intravenous bolus injection into the venous line of the dialysis circuit at the end of each dialysis.
  Arms: 12-weeks double-blind period-QLG2198; 14-weeks open-label period following the double-blind period- QLG2198
Drug: Placebo — Participants receive Placebo three times a week (0,5 micrograms/kg dry body weight). Placebo is administered by intravenous bolus injection into the venous line of the dialysis circuit at the end of each dialysis
  Arms: 12-weeks double-blind period- placebo

SUMMARY:
This a multicentre study that consists of a 12-week double-blind period, and a 14-week open-label extension period and a 1-week follow-up period.

DETAILED DESCRIPTION:
Total study duration for a single subject is 31 to 32 weeks with a 4-week screening period, a 12-week double-blind period, a 14-week open-label extension period, and a 1-week follow-up period.

QLG2198 will be administered in the double-blind and open-label period 3 times a week at the end of each dialysis session. The total dose of the investigational product will be determined based on the subject's prescription dry body weight.

The primary objective of the study is:

To evaluate the efficacy and safety of QLG2198 0.5 μg/kg compared to placebo in reducing the intensity of itch in HD subjects with moderate-to-severe pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic kidney disease (CKD) on HD 3 times weekly for ≥12 weeks prior to screening who can continue HD without changing its frequency or method
* If female, is not pregnant, or nursing.
* agrees not to donate sperm or egg after the first dose of investigational product administration until 7 days after the last dose of investigational product, and agrees to use contraceptive method from heterosexual intercourse during the study until 7 days after the last dose of investigational product.
* Subjects with a prescription dry body weight between 40 and 100 kg

Exclusion Criteria:

* Planned to receive a kidney transplant during the study.
* Has localised itch restricted to the palms of the hands.
* Has pruritus only during the dialysis session
* Subjects with severe hepatic impairment (Child-Pugh Class C) or concurrent hepatic cirrhosis.
* Subject is receiving ongoing ultraviolet treatment .
* Subjects with concurrent malignancy except excised basal cell or squamous cell carcinoma of the skin, or carcinoma in situ that has been excised or resected completely.
* Known or suspected history of alcohol or drug abuse/dependence within 12 months prior to screening.
* New or change of treatment received for itch within 2 weeks prior to screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-02-21 (Estimated); Study Completion 2025-08-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the weekly mean of the Worst Itch Numeric Rating Scale (WI-NRS) score | Week 4 of double-blind period
  The degree of the most intense itching within a day will be assessed using Worst Itch Numeric Rating Scale (WI-NRS) scores.patients will be asked to indicate the intensity of the worst itching they experienced over the past 24 hours by marking one of 11 numbers, from 0 to 10, that best describes it, where "0" is labeled with the anchor phrase "no itching" and "10" is labeled "worst itching imaginable."

SECONDARY OUTCOMES:
Proportion of subjects achieving ≥3-point improvement from baseline with respect to the weekly mean of the WI-NRS | Week 4 、Week 8、 Week 12 of double-blind period
  The degree of the most intense itching within a day will be assessed using Worst Itch Numeric Rating Scale (WI-NRS) scores.
Proportion of subjects achieving ≥4-point improvement from baseline with respect to the weekly mean of the WI-NRS | Week 4 、Week 8、 Week 12 of double-blind period
  The degree of the most intense itching within a day will be assessed using Worst Itch Numeric Rating Scale (WI-NRS) scores.
Change from baseline in itch-related Quality of Life (QoL) assessed by the 5-D itch scale total score | Week 4 、Week 8、Week 12 of double-blind period,Week 4 、Week 8、Week 12 、Week 15 of open-label extension period
  The 5-D itch scale is a questionnaire where patients assess the 5 dimensions of itch (degree, duration, direction, disability, and distribution).The total score is the sum of the numeric value of each answered question.
Change from baseline in itch-related QoL assessed by the Skindex-10 scale total score | Week 4 、Week 8、 Week 12 of double-blind period,Week 4 、Week 8、Week 12 、Week 15 of open-label extension period
  The Skindex-10 scale is a questionnaire that measures QoL in relationship to the itch intensity.Patients are asked to mark 1 of 7 boxes numbered from 0(labeled with the anchor phrase "never bothered") to 6 (labeled as "always bothered") for each of the 10 questions describing how often they have been bothered by their itch and its impact over the past week. The total score is the sum of the numeric value of each answered question. The total score is subdivided into 3 domain scores, which are sums of the scores of the following questions: disease domain (questions 1 to 3),mood/emotional distress domain (questions 4 to 6), and social functioning domain (questions 7 to 10).
Patient Global Impression of Change | End of double-blind period, week 12
  The Patient Global Impression of Change is a questionnaire that assesses the change in itch compared to the itch at the start of the study.The scale has only 1 item, and the patient is asked to mark the category that best describes the change in itch ranging from "Very Much Improved" to"Very Much Worse"

CONTACTS AND LOCATIONS:
Overall Officials: Zuo Li, Principal Investigator — Peking University People's Hospital; Wang Rong, Principal Investigator — Shandong Provincial Hospital
Locations (3):
- China (3):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Shandong Provincial Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No